CLINICAL TRIAL: NCT01862172
Title: FOCAL CORTICAL ATROPHY AFTER MYOCARDIAL INTERNAL CAPSULE: CORRELATION FRACTION ANISOTROPY BEAM PYRAMID AND DISABILITY
Brief Title: Focal Cortical Atrophy After Myocardial Internal Capsule
Acronym: ACFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12 486 03; HAO 2012 (Other: University Hospital of Toulouse)
Record Dates: First submitted 2013-04-29; First posted 2013-05-24 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Ischemic Stroke
Keywords: Cortical focal atrophy; Stroke; Internal capsule; Corticospinal tract; Wallerian degeneration; Primary motor area.
MeSH Terms: conditions — Ischemic Stroke; Stroke; Wallerian Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- additional MRI (Other)
  Interventions: Other: Additional MRI

INTERVENTIONS:
Other: Additional MRI

SUMMARY:
Primary purpose of the trial is to demonstrate the arisen of focal cortical atrophy, localized in the ipsilateral primary motor area, measured in mm, three months after infarction of internal capsule.

The patient is compared to himself between day zero to ten and three months.

The study hypotheses are:

* A focal cortical atrophy of the ipsilesional primary motor area occurs after cerebral infarction of the internal capsule. It is measurable accurately and reproducibly by MRI at three months. Other brain areas within the voluntary motor system will also be explored (supplementary motor area, pre motor area).
* This atrophy is correlated with achievement of pyramidal tract, assessed by the fractional anisotropy of its fibers.
* This atrophy is correlated with disability at three months, assessed by Rankin score.

DETAILED DESCRIPTION:
Twenty-two patients with ischemic stroke, subcortical, involving the internal capsule, will be included.

Each patient will be compared to himself, on day zero to ten and three months.

An MRI will be performed between day zero and ten, then three months of infarction sequences with traditional threeD enabling acquisition and tractography and The measurement of cortical thickness is in mm The measurement of fractional anisotropy of the pyramidal tract A clinical evaluation will be done between Day zero and Day ten then three months, using a neurological score (NIHSS), a score of functional disability (Rankin) and more analytical and sensitive tests such as dynamometer, the Finger Tapping test and test new plugs.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 18 to 90 years old.
* Subcortical stroke
* Achievement of the internal capsule, according to MRI
* Ability to perform MRI within 10 days after the onset of symptoms
* NIHSS over or equal 2 and < 20
* Rankin Score over or equal 1 and ≤ 5
* Written informed consent after information about the protocol, from patients or reliable person if patient is in incapacity to sign
* Affiliation to a social security scheme

Exclusion Criteria:

* Pregnant or nursing women
* Other cerebral lesion, concomitant or preexisting
* Concomitant disease causing unfavorable prognosis within 3 months after inclusion
* pre-existing psychiatric illness
* Alcoholism or other chronic intoxication
* Cortical localization of the infarction
* Patient in a coma, who cannot be examined and evaluated
* Patient intubated, ventilated, sedated
* Cerebral hemorrhage, intra-parenchymal and / or subarachnoid
* Persons protected by law (guardianship, curators and judicial protection)
* Contraindications to magnetic resonance examination: pacemaker, metal implants, neurostimulators, Clips neurosurgical wire sutures, staples, metal heart valves, ventricular bypass valve, metal workers, foreign eye, shrapnel, bullet , cochlear implants

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Decrease of cortical thickness | 3 months after infarction of corticospinal tract, in the ipsilateral primary motor area.
  Decrease of cortical thickness in the ipsilateral primary motor area, after infarction of corticospinal tract at 3 months.

SECONDARY OUTCOMES:
Calculation of fractional anisotropy | 3 months after infarction of corticospinal tract
  Calculation of fractional anisotropy will be done through the sequence MRI tractography to D0-D10 and 3 months
Disability | at 3 months
  The disability at 3 months will be evaluated with the Rankin score

CONTACTS AND LOCATIONS:
Overall Officials: François CHOLLET, PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, Midi-Pyrenees, France

REFERENCES:
- [Background] Ashburner J, Friston K. Multimodal image coregistration and partitioning--a unified framework. Neuroimage. 1997 Oct;6(3):209-17. doi: 10.1006/nimg.1997.0290. PMID 9344825
- [Background] Bloch I Fuzzy spatial relationships for image processing and interpretation: a review. Image Vis Comput 2004;23:89-110.
- [Background] Kolb B. Recovery from early cortical damage in rats. I. Differential behavioral and anatomical effects of frontal lesions at different ages of neural maturation. Behav Brain Res. 1987 Sep;25(3):205-20. doi: 10.1016/0166-4328(87)90069-6. PMID 3689568
- [Background] Stinear CM, Barber PA, Smale PR, Coxon JP, Fleming MK, Byblow WD. Functional potential in chronic stroke patients depends on corticospinal tract integrity. Brain. 2007 Jan;130(Pt 1):170-80. doi: 10.1093/brain/awl333. PMID 17148468
- [Background] Preul C, Lohmann G, Hund-Georgiadis M, Guthke T, von Cramon DY. Morphometry demonstrates loss of cortical thickness in cerebral microangiopathy. J Neurol. 2005 Apr;252(4):441-7. doi: 10.1007/s00415-005-0671-9. Epub 2005 Feb 23. PMID 15726260
- [Background] Tur C, Penny S, Khaleeli Z, Altmann DR, Cipolotti L, Ron M, Thompson AJ, Ciccarelli O. Grey matter damage and overall cognitive impairment in primary progressive multiple sclerosis. Mult Scler. 2011 Nov;17(11):1324-32. doi: 10.1177/1352458511410341. Epub 2011 Jul 29. PMID 21803874
- [Background] DeCarli C, Massaro J, Harvey D, Hald J, Tullberg M, Au R, Beiser A, D'Agostino R, Wolf PA. Measures of brain morphology and infarction in the framingham heart study: establishing what is normal. Neurobiol Aging. 2005 Apr;26(4):491-510. doi: 10.1016/j.neurobiolaging.2004.05.004. PMID 15653178
- [Background] Fein G, Di Sclafani V, Tanabe J, Cardenas V, Weiner MW, Jagust WJ, Reed BR, Norman D, Schuff N, Kusdra L, Greenfield T, Chui H. Hippocampal and cortical atrophy predict dementia in subcortical ischemic vascular disease. Neurology. 2000 Dec 12;55(11):1626-35. doi: 10.1212/wnl.55.11.1626. PMID 11113215
- [Background] Gerloff C, Bushara K, Sailer A, Wassermann EM, Chen R, Matsuoka T, Waldvogel D, Wittenberg GF, Ishii K, Cohen LG, Hallett M. Multimodal imaging of brain reorganization in motor areas of the contralesional hemisphere of well recovered patients after capsular stroke. Brain. 2006 Mar;129(Pt 3):791-808. doi: 10.1093/brain/awh713. Epub 2005 Dec 19. PMID 16364955
- [Background] Green HA, Pena A, Price CJ, Warburton EA, Pickard JD, Carpenter TA, Gillard JH. Increased anisotropy in acute stroke: a possible explanation. Stroke. 2002 Jun;33(6):1517-21. doi: 10.1161/01.str.0000016973.80180.7b. PMID 12052984
- [Background] Grefkes C, Eickhoff SB, Nowak DA, Dafotakis M, Fink GR. Dynamic intra- and interhemispheric interactions during unilateral and bilateral hand movements assessed with fMRI and DCM. Neuroimage. 2008 Jul 15;41(4):1382-94. doi: 10.1016/j.neuroimage.2008.03.048. Epub 2008 Apr 8. PMID 18486490
- [Background] Goldman AL, Pezawas L, Mattay VS, Fischl B, Verchinski BA, Chen Q, Weinberger DR, Meyer-Lindenberg A. Widespread reductions of cortical thickness in schizophrenia and spectrum disorders and evidence of heritability. Arch Gen Psychiatry. 2009 May;66(5):467-77. doi: 10.1001/archgenpsychiatry.2009.24. PMID 19414706
- [Background] Jones SE, Buchbinder BR, Aharon I. Three-dimensional mapping of cortical thickness using Laplace's equation. Hum Brain Mapp. 2000 Sep;11(1):12-32. doi: 10.1002/1097-0193(200009)11:13.0.co;2-k. PMID 10997850
- [Background] Schaechter JD, Moore CI, Connell BD, Rosen BR, Dijkhuizen RM. Structural and functional plasticity in the somatosensory cortex of chronic stroke patients. Brain. 2006 Oct;129(Pt 10):2722-33. doi: 10.1093/brain/awl214. Epub 2006 Aug 18. PMID 16921177
- [Background] Puig J, Pedraza S, Blasco G, Daunis-I-Estadella J, Prats A, Prados F, Boada I, Castellanos M, Sanchez-Gonzalez J, Remollo S, Laguillo G, Quiles AM, Gomez E, Serena J. Wallerian degeneration in the corticospinal tract evaluated by diffusion tensor imaging correlates with motor deficit 30 days after middle cerebral artery ischemic stroke. AJNR Am J Neuroradiol. 2010 Aug;31(7):1324-30. doi: 10.3174/ajnr.A2038. Epub 2010 Mar 18. PMID 20299434
- [Background] Kraemer M, Schormann T, Hagemann G, Qi B, Witte OW, Seitz RJ. Delayed shrinkage of the brain after ischemic stroke: preliminary observations with voxel-guided morphometry. J Neuroimaging. 2004 Jul;14(3):265-72. doi: 10.1177/1051228404264950. PMID 15228769
- [Background] Kunimatsu A, Aoki S, Masutani Y, Abe O, Mori H, Ohtomo K. Three-dimensional white matter tractography by diffusion tensor imaging in ischaemic stroke involving the corticospinal tract. Neuroradiology. 2003 Aug;45(8):532-5. doi: 10.1007/s00234-003-0974-4. Epub 2003 Jul 11. PMID 12856090
- [Background] Konishi J, Yamada K, Kizu O, Ito H, Sugimura K, Yoshikawa K, Nakagawa M, Nishimura T. MR tractography for the evaluation of functional recovery from lenticulostriate infarcts. Neurology. 2005 Jan 11;64(1):108-13. doi: 10.1212/01.WNL.0000148477.65273.0C. PMID 15642912
- [Background] Lauretani F, Saccavini M, Zaccaria B, Agosti M, Zampolini M, Franceschini M; ICR2 Group. Rehabilitation in patients affected by different types of stroke. A one-year follow-up study. Eur J Phys Rehabil Med. 2010 Dec;46(4):511-6. Epub 2010 Apr 23. PMID 20414185
- [Background] Radlinska B, Ghinani S, Leppert IR, Minuk J, Pike GB, Thiel A. Diffusion tensor imaging, permanent pyramidal tract damage, and outcome in subcortical stroke. Neurology. 2010 Sep 21;75(12):1048-54. doi: 10.1212/WNL.0b013e3181f39aa0. PMID 20855848
- [Background] Lerch JP, Evans AC. Cortical thickness analysis examined through power analysis and a population simulation. Neuroimage. 2005 Jan 1;24(1):163-73. doi: 10.1016/j.neuroimage.2004.07.045. PMID 15588607
- [Background] Gauthier LV, Taub E, Mark VW, Barghi A, Uswatte G. Atrophy of spared gray matter tissue predicts poorer motor recovery and rehabilitation response in chronic stroke. Stroke. 2012 Feb;43(2):453-7. doi: 10.1161/STROKEAHA.111.633255. Epub 2011 Nov 17. PMID 22096036
- [Background] Mark VW, Taub E, Perkins C, Gauthier L, Uswatte G. MRI infarction load and CI therapy outcomes for chronic post-stroke hemiparesis. Restor Neurol Neurosci. 2008;26(1):13-33. PMID 18431003
- [Background] Calabrese M, Agosta F, Rinaldi F, Mattisi I, Grossi P, Favaretto A, Atzori M, Bernardi V, Barachino L, Rinaldi L, Perini P, Gallo P, Filippi M. Cortical lesions and atrophy associated with cognitive impairment in relapsing-remitting multiple sclerosis. Arch Neurol. 2009 Sep;66(9):1144-50. doi: 10.1001/archneurol.2009.174. PMID 19752305
- [Background] Mori S, Crain BJ, Chacko VP, van Zijl PC. Three-dimensional tracking of axonal projections in the brain by magnetic resonance imaging. Ann Neurol. 1999 Feb;45(2):265-9. doi: 10.1002/1531-8249(199902)45:23.0.co;2-3. PMID 9989633
- [Background] Querbes O, Aubry F, Pariente J, Lotterie JA, Demonet JF, Duret V, Puel M, Berry I, Fort JC, Celsis P; Alzheimer's Disease Neuroimaging Initiative. Early diagnosis of Alzheimer's disease using cortical thickness: impact of cognitive reserve. Brain. 2009 Aug;132(Pt 8):2036-47. doi: 10.1093/brain/awp105. Epub 2009 May 12. PMID 19439419
- [Background] Pierpaoli C, Basser PJ. Toward a quantitative assessment of diffusion anisotropy. Magn Reson Med. 1996 Dec;36(6):893-906. doi: 10.1002/mrm.1910360612. PMID 8946355
- [Background] Swartz RH, Stuss DT, Gao F, Black SE. Independent cognitive effects of atrophy and diffuse subcortical and thalamico-cortical cerebrovascular disease in dementia. Stroke. 2008 Mar;39(3):822-30. doi: 10.1161/STROKEAHA.107.491936. Epub 2008 Feb 7. PMID 18258840
- [Background] Ross ED. Localization of the pyramidal tract in the internal capsule by whole brain dissection. Neurology. 1980 Jan;30(1):59-64. doi: 10.1212/wnl.30.1.59. PMID 7188635
- [Background] Schormann T, Kraemer M. Voxel-guided morphometry ("VGM") and application to stroke. IEEE Trans Med Imaging. 2003 Jan;22(1):62-74. doi: 10.1109/TMI.2002.806571. PMID 12703760
- [Background] Thomalla G, Glauche V, Koch MA, Beaulieu C, Weiller C, Rother J. Diffusion tensor imaging detects early Wallerian degeneration of the pyramidal tract after ischemic stroke. Neuroimage. 2004 Aug;22(4):1767-74. doi: 10.1016/j.neuroimage.2004.03.041. PMID 15275932
- [Background] Wang LE, Fink GR, Diekhoff S, Rehme AK, Eickhoff SB, Grefkes C. Noradrenergic enhancement improves motor network connectivity in stroke patients. Ann Neurol. 2011 Feb;69(2):375-88. doi: 10.1002/ana.22237. Epub 2010 Dec 28. PMID 21387380
- [Background] Xue R, van Zijl PC, Crain BJ, Solaiyappan M, Mori S. In vivo three-dimensional reconstruction of rat brain axonal projections by diffusion tensor imaging. Magn Reson Med. 1999 Dec;42(6):1123-7. doi: 10.1002/(sici)1522-2594(199912)42:63.0.co;2-h. PMID 10571934
- [Background] Yagishita A, Nakano I, Oda M, Hirano A. Location of the corticospinal tract in the internal capsule at MR imaging. Radiology. 1994 May;191(2):455-60. doi: 10.1148/radiology.191.2.8153321.
- [Background] Yang Q, Tress BM, Barber PA, Desmond PM, Darby DG, Gerraty RP, Li T, Davis SM. Serial study of apparent diffusion coefficient and anisotropy in patients with acute stroke. Stroke. 1999 Nov;30(11):2382-90. doi: 10.1161/01.str.30.11.2382. PMID 10548675
- [Background] Zhu LL, Lindenberg R, Alexander MP, Schlaug G. Lesion load of the corticospinal tract predicts motor impairment in chronic stroke. Stroke. 2010 May;41(5):910-5. doi: 10.1161/STROKEAHA.109.577023. Epub 2010 Apr 8. PMID 20378864
- [Derived] Loubinoux I, Lafuma M, Rigal J, Colitti N, Albucher JF, Raposo N, Planton M, Olivot JM, Chollet F. Diffusion tensor imaging and gray matter volumetry to evaluate cerebral remodeling processes after a pure motor stroke: a longitudinal study. J Neurol. 2024 Oct;271(10):6876-6887. doi: 10.1007/s00415-024-12648-y. Epub 2024 Sep 3. PMID 39223359